CLINICAL TRIAL: NCT01211145
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, 4-Armed Parallel Group Study to Evaluate the Efficacy of Zolmitriptan 0.5-, 2.5- and 5-mg Nasal Spray in the Treatment of Acute Migraine Headache in Adolescents
Brief Title: Zomig - Treatment of Acute Migraine Headache in Adolescents
Acronym: TEENZ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1220C00001
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Migraine Headache
Keywords: Migraine; Headache; Pain; Efficacy; Adolescents
MeSH Terms: conditions — Migraine Disorders; Headache; Pain | interventions — zolmitriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): ZOMIG 0.5 mg
  Interventions: Drug: Zolmitriptan
- 3 (Experimental): ZOMIG 2.5 mg
  Interventions: Drug: Zolmitriptan
- 4 (Experimental): ZOMIG 5.0 mg
  Interventions: Drug: Zolmitriptan

INTERVENTIONS:
Drug: Placebo — Placebo nasal spray
  Arms: 1
Drug: Zolmitriptan — 0.5 mg nasal spray
  Other Names: Zomig® Nasal Spray
  Arms: 2
Drug: Zolmitriptan — 2.5 mg nasal spray
  Other Names: Zomig® Nasal Spray
  Arms: 3
Drug: Zolmitriptan — 5.0 mg nasal spray
  Other Names: Zomig® Nasal Spray
  Arms: 4

SUMMARY:
The purpose of this study is to investigate if Zomig® Nasal Spray will help children (age 12-17 years) with migraine headaches feel better. This will be done by comparing 3 different doses of Zomig Nasal Spray with placebo nasal spray (inactive treatment).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent by parent or legal guardian, and written assent provided by patient prior to any study specific procedures.
* Established diagnosis of migraine.
* History of a minimum of 2 migraine attacks (moderately or severely disabling)per month.

Exclusion Criteria:

* Any medical condition that may put the patient at increased risk with exposure to zolmitriptan or that may interfere with the safety or efficacy assessments.
* A history of basilar, ophthalmoplegic, or hemiplegic migraine headache or any potentially serious neurological condition that is associated with headache.
* Have had an unacceptable adverse experience following previous use of any 5HT1B/1D agonist drug.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1653 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohini Chitra, Study Director — AZ Pharmaceuticals, US; Paul Winner, Principal Investigator — Children's Hospital of The King's Daughters
Locations (74):
- United States (46):
  - Research Site, Phoenix, Arizona
  - Research Site, Fresno, California
  - Research Site, Fullerton, California
  - Research Site, Newport Beach, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Centennial, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Thornton, Colorado
  - Research Site, Fairfield, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Hallandale, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, North Palm Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Owensboro, Kentucky
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Plymouth, Minnesota
  - Research Site, Ocean Springs, Mississippi
  - Research Site, Olive Branch, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, The Bronx, New York
  - Research Site, Cary, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Indiana, Pennsylvania
  - Research Site, Jackson, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Spring, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, South Jordan, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Middleton, Wisconsin
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Mikkeli
  - Research Site, Turku
- Hungary (9):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyula
  - Research Site, Miskolc
  - Research Site, Nagykanizsa
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Sopron
  - Research Site, Szekszárd
- Latvia (2):
  - Research Site, Riga
  - Research Site, Valmiera
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Kielce
  - Research Site, Olsztyn
  - Research Site, Poznan
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Novi Sad
- Slovakia (3):
  - Research Site, Dolný Kubín
  - Research Site, Nitra
  - Research Site, Zvolen

REFERENCES:
- See also: D1220C00001 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1740&filename=D1220C00001_CSR_Synopsis.pdf
- See also: D1220C00001 Revised CSP 3 Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1740&filename=D1220C00001%20Revised%20CSP%203%20No%20Futility_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted between 7 October 2010 and 31 October 2013.
Pre-assignment Details: The study had a 30 day run-in period and up to a 10-week double-blind treatment period. Patients were randomized to receive ZOMIG nasal spray 0.5, 2.5, 5.0 mg, or matching placebo spray to treat a migraine headache. 1653 patients were enrolled, 798 were randomized.
Groups:
- Placebo: Placebo to ZOMIG nasal spray
- ZOMIG 0.5 mg; ZOMIG 2.5 mg; ZOMIG 5 mg: ZOMIG nasal spray
Period: Overall Study
Arm/Group | Placebo | ZOMIG 0.5 mg | ZOMIG 2.5 mg | ZOMIG 5 mg
Started | 296 | 115 | 99 | 288
Completed | 270 (1 patient was not counted as completed or discontinued due to incomplete information (N=270-1=269).) | 98 | 86 | 268
Not Completed | 26 | 17 | 13 | 20
Not completed — Reason not specified | 3 | 2 | 2 | 1
Not completed — Lost to Follow-up | 3 | 2 | 1 | 2
Not completed — Study-specific withdrawal criteria | 1 | 0 | 0 | 0
Not completed — Severe noncompliance to protocol | 1 | 0 | 0 | 0
Not completed — Eligibility criteria not fulfilled | 16 | 12 | 10 | 15
Not completed — Patient decision | 2 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ZOMIG 0.5 mg | ZOMIG 2.5 mg | ZOMIG 5 mg | Total
Number analyzed (Participants) | 296 | 115 | 99 | 288 | 798
Age, Continuous [Mean (Standard Deviation); unit: Years] — All randomized patients
  Years | 14.3 (1.67) | 14.5 (1.72) | 14.6 (1.77) | 14.5 (1.67) | 14.4 (1.69)
Sex: Female, Male [Count of Participants; unit: Participants] — All randomized patients
  Participants
    Female | 188 | 71 | 62 | 172 | 493
    Male | 108 | 44 | 37 | 116 | 305

OUTCOME MEASURES:

1. Primary Outcome: Pain-free Status at 2 Hours Post-treatment
Time Frame: 2 hours post-treatment.
Population: Full analysis set (last observation carried forward)
Measure: Number; unit: Participants
Arm/Group | Placebo | ZOMIG 0.5 mg | ZOMIG 2.5 mg | ZOMIG 5 mg
Number analyzed (Participants) | 253 | 91 | 81 | 229
Participants
  Yes | 42 | 20 | 20 | 68
  No | 211 | 71 | 61 | 161
Statistical Analysis 1: Comparison: Placebo vs ZOMIG 0.5 mg; Test type: Superiority or Other; p = .312, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.75 to 2.50] — ZOMIG 0.5 mg/Placebo
Statistical Analysis 2: Comparison: Placebo vs ZOMIG 2.5 mg; Test type: Superiority or Other; p = .071, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.95 to 3.26] — ZOMIG 2.5 mg/Placebo
Statistical Analysis 3: Comparison: Placebo vs ZOMIG 5 mg; Test type: Superiority or Other; p < .001, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 2.18, 95% CI 2-sided [1.40 to 3.39] — ZOMIG 5.0 mg/Placebo

2. Secondary Outcome: Pain-free Status at 24 Hours Post-treatment
Time Frame: 24 hours post-treatment
Population: Full analysis set (observed case)
Measure: Number; unit: Participants
Arm/Group | Placebo | ZOMIG 0.5 mg | ZOMIG 2.5 mg | ZOMIG 5 mg
Number analyzed (Participants) | 251 | 91 | 80 | 227
Participants
  Yes | 155 | 59 | 60 | 155
  No | 96 | 32 | 20 | 72
Statistical Analysis 1: Comparison: Placebo vs ZOMIG 0.5 mg; Test type: Superiority or Other; p = .575, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.70 to 1.91] — ZOMIG 0.5 mg/Placebo
Statistical Analysis 2: Comparison: Placebo vs ZOMIG 2.5 mg; Test type: Superiority or Other; p = .032, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.06 to 3.31] — ZOMIG 2.5 mg/Placebo
Statistical Analysis 3: Comparison: Placebo vs ZOMIG 5 mg; Test type: Superiority or Other; p = .137, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.91 to 1.95] — ZOMIG 5.0 mg/Placebo

3. Secondary Outcome: Headache Response at 2 Hours Post-treatment
Description: Headache response is a binary response variable derived from the headache intensities recorded in the patient diary. Headache response is defined as a reduction in headache pain intensity from severe or moderate to mild or none with no use of rescue medication prior to the assessment.
Time Frame: 2 hours post-treatment
Population: Full analysis set (last observation carried forward)
Measure: Number; unit: Participants
Arm/Group | Placebo | ZOMIG 0.5 mg | ZOMIG 2.5 mg | ZOMIG 5 mg
Number analyzed (Participants) | 253 | 91 | 81 | 229
Participants
  Yes | 99 | 40 | 43 | 116
  No | 154 | 51 | 38 | 113
Statistical Analysis 1: Comparison: Placebo vs ZOMIG 0.5 mg; Test type: Superiority or Other; p = .458, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.74 to 1.96] — ZOMIG 0.5 mg/Placebo
Statistical Analysis 2: Comparison: Placebo vs ZOMIG 2.5 mg; Test type: Superiority or Other; p = .021, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.09 to 3.03] — ZOMIG 2.5 mg/Placebo
Statistical Analysis 3: Comparison: Placebo vs ZOMIG 5 mg; Test type: Superiority or Other; p = .010, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.12 to 2.32] — ZOMIG 5.0 mg/Placebo

4. Secondary Outcome: Headache Response at 24 Hours Post-treatment
Description: as for outcome 3
Time Frame: 24 hours post-treatment
Population: Full analysis set (observed case)
Measure: Number; unit: Participants
Arm/Group | Placebo | ZOMIG 0.5 mg | ZOMIG 2.5 mg | ZOMIG 5 mg
Number analyzed (Participants) | 251 | 91 | 80 | 227
Participants
  Yes | 170 | 63 | 61 | 168
  No | 81 | 28 | 19 | 59
Statistical Analysis 1: Comparison: Placebo vs ZOMIG 0.5 mg; Test type: Superiority or Other; p = .753, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.64 to 1.84] — ZOMIG 0.5 mg/Placebo
Statistical Analysis 2: Comparison: Placebo vs ZOMIG 2.5 mg; Test type: Superiority or Other; p = .145, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.86 to 2.79] — ZOMIG 2.5 mg/Placebo
Statistical Analysis 3: Comparison: Placebo vs ZOMIG 5 mg; Test type: Superiority or Other; p = .127, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.91 to 2.04] — ZOMIG 5.0 mg/Placebo

5. Secondary Outcome: Sustained Headache Response at 2 Hours
Description: Sustained headache response at 2 hours is a binary response variable derived from the headache intensities recorded in the patient diary. Sustained headache response is defined as a reduction in migraine headache pain intensity from severe or moderate to mild or none a 1 hr. which is then maintained (without a return to moderate or severe pain) at 2 hrs. with no use of rescue medication prior to the 2 hr. assessment.
Time Frame: Up to 2 hours post-treatment
Population: Full analysis set (observed case)
Measure: Number; unit: Participants
Arm/Group | Placebo | ZOMIG 0.5 mg | ZOMIG 2.5 mg | ZOMIG 5 mg
Number analyzed (Participants) | 251 | 91 | 81 | 224
Participants
  Yes | 59 | 27 | 27 | 66
  No | 192 | 64 | 54 | 158
Statistical Analysis 1: Comparison: Placebo vs ZOMIG 0.5 mg; Test type: Superiority or Other; p = .274, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.79 to 2.32] — ZOMIG 0.5 mg/Placebo
Statistical Analysis 2: Comparison: Placebo vs ZOMIG 2.5 mg; Test type: Superiority or Other; p = .067, Regression, Logistic — Unadjusted; Odds Ratio, log = 1.67, 95% CI 2-sided [0.96 to 2.91] — ZOMIG 2.5 mg/Placebo
Statistical Analysis 3: Comparison: Placebo vs ZOMIG 5 mg; Test type: Superiority or Other; p = .127, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.91 to 2.08] — ZOMIG 5.0 mg/Placebo

6. Secondary Outcome: Use of Rescue Medication During the First 24 Hours After Treatment
Time Frame: 24 hours post-treatment.
Population: Full analysis set (observed cases)
Measure: Number; unit: Participants
Arm/Group | Placebo | ZOMIG 0.5 mg | ZOMIG 2.5 mg | ZOMIG 5 mg
Number analyzed (Participants) | 253 | 91 | 81 | 231
Participants
  Yes | 80 | 22 | 18 | 47
  No | 173 | 69 | 63 | 184
Statistical Analysis 1: Comparison: Placebo vs ZOMIG 0.5 mg; Test type: Superiority or Other; p = .153, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.38 to 1.16] — ZOMIG 0.5 mg/Placebo
Statistical Analysis 2: Comparison: Placebo vs ZOMIG 2.5 mg; Test type: Superiority or Other; p = .087, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.33 to 1.08] — ZOMIG 2.5 mg/Placebo
Statistical Analysis 3: Comparison: Placebo vs ZOMIG 5 mg; Test type: Superiority or Other; p = .004, Regression, Logistic — Unadjusted; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.36 to 0.83] — ZOMIG 5.0 mg/Placebo

ADVERSE EVENTS:
Description: Safety Analysis Set (Number of Patients at Risk: Placebo=253; ZOMIG 0.5 mg=92; ZOMIG 2.5 mg=81; ZOMIG 5 mg=231)
Arm/Group | Placebo | ZOMIG 0.5 mg | ZOMIG 2.5 mg | ZOMIG 5 mg
Serious Adverse Events (participants affected / at risk) | 0/253 | 0/92 | 0/81 | 0/231
Other Adverse Events (participants affected / at risk) | 25/253 | 14/92 | 9/81 | 59/231
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=253) | ZOMIG 0.5 mg (N=92) | ZOMIG 2.5 mg (N=81) | ZOMIG 5 mg (N=231)
Dysgeusia (Nervous system disorders) | 3 (3) | 6 (6) | 5 (5) | 29 (29)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 6 (6)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 2 (2) | 7 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 7 (7)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Bradykinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Administration related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other